CLINICAL TRIAL: NCT05790915
Title: Impact of Interventions on Admission SOFA Score on Clinical Outcomes of Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, ICU Assistant Physician, Hospital Sao Domingos
Other Study IDs: HSD 2023 1
Record Dates: First submitted 2023-02-21; First posted 2023-03-30 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Critically Ill Patients
Keywords: SOFA Score; Delta SOFA; Critically ill patients; Interventions; Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with SOFA score < 2 at admission. No intervention
- Group 2: Patients with SOFA score equal to or > 2 on admission and who improved after 48 hours of treatment.
  Intervention focused on identified organ dysfunction(s)
  Interventions: Combination Product: Standardized interventions
- Group 3: Patients with SOFA score equal to or > 2 on admission and who did not improve after 48 hours of treatment.
  Intervention focused on identified organ dysfunction(s)
  Interventions: Combination Product: Standardized interventions

INTERVENTIONS:
Combination Product: Standardized interventions — Standardized interventions according organ dysfunction
  Groups: Group 2; Group 3

SUMMARY:
Introduction: The SOFA score (Sequential Organ Function Assessment) and its derived measures, such as the Delta SOFA, are used worldwide to determine the severity and prognosis of critically ill patients.

Objectives: The primary objective of this study was to assess the impact of standardized interventions on the six organ dysfunctions of SOFA score on outcomes of critically ill patients through the 48-hour delta SOFA with evaluation of the effectiveness of the interventions performed. Result will be correlated with the 28-day mortality.

The secondary outcome measures comprised the evaluation of standardized interventions on ICU and hospital length of stay; vasopressor-free and ventilator-free days within the 28 days following ICU admission, through the effectiveness of interventions performed Uni and multivariate statistical analysis will be used to determine organ failures associated to outcome.

DETAILED DESCRIPTION:
This prospective, observational cohort study will include patients admitted to a medical ICU (12 beds), a surgical ICU (13 beds), and a high complexity surgical and trauma ICU (12 beds). of a tertiary hospital from August 01, 2023 to January31, 2024. The trial will include all patients aged above 18 years, admitted to the ICU for at least 3 days. Patients will be excluded for the following reasons: if they are pregnant, moribund and patients readmitted to the ICU in the same hospital admission.

For the patients who met the inclusion criteria, we will collect the demographic data regarding the age, gender, the admission category (medical or surgical), the primary admission diagnosis, the simplified acute physiology score III (SAPS 3), admission sequential organ failure assessment (SOFA) and 48-hour SOFA.

Whenever the admission SOFA score is ≥ 2, the result will be presented to the attending physician who will establish in the therapeutic plan the interventions for each of the dysfunctions identified according to a standardized intervention protocol (Table 1). After 48 hours, a new SOFA score is determined, while the prospective clinical surveillance team simultaneously identify if the interventions proposed by the protocol for each of the organ dysfunctions were effectively implemented.

Three groups of patients will be identified based on their SOFA scores at admission and the 48-hour delta SOFA values: those with an admission SOFA score < 2 (Group1), those with an admission SOFA score ≥ 2 whose delta SOFA reflected improvement at the end of 48 hours after admission (SOFA after 48 hours < SOFA on admission) (Group 2, n= ) and finally, those with an admission SOFA score ≥ 2 whose SOFA score increased or remained unchanged at the end of 48 hours postadmission (SOFA after 48 hours ≥ admission SOFA) (Group 3, n= ). The effectiveness of the interventions on organic disfunction will be evaluated in the groups 2 and 3 through the formula:

Number of patients with an organic disfunction and effective intervention / Number of patients with that organic dysfunction X 100

Results will be correlated with 28-day mortality.

Table 1. SOFA standardized protocol

1. Respiratory Protective mechanical ventilation; mechanical power < 16 NIV Prevention of P-SILI: ROX and HACOR index
2. Hemodynamic SOSD protocol; Pressoric target; Lactate clearance
3. Neurologic Image; EEG; Sedation goals
4. Hematologic Basic disease approach; drugs; DDAVP use; platelet transfusion
5. Renal Avoid nephrotoxicity; Avoid hypotension
6. Hepatic Avoid hepatotoxic drugs; basic disease approach.

NIV, Non-invasive ventilation; P-SILI, patient self-inflicted lung injury; ROX, ratio of oxygen saturation index; HACOR, Heart rate, acidosis, consciousness oxygenatrion and respiratory rate; SOSD, salvage, optimization, stabilization and de-escalation; DDAVP, 1-desamino-8-d-arginine-vasopresssin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 18 years,
* Lenght of ICU stay of at least 3 days.

Exclusion Criteria:

* Pregnant patients
* End-of-life
* Patients readmitted to the ICU in the same hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to a medical ICU, a Surgical ICU and a High complexity surgical and trauma ICU in the period from April 01, 2023 to March 31, 2024 and lenght of stay of at least 3 days.
Sampling Method: Probability Sample
Enrollment: 849 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Impact of standardized interventions in respiratory dysfunction on 48-hour delta SOFA with evaluation of the effectiveness of the interventions performed. | 48 hours
  Lung protective ventilation: Tidal volume = 6 ml/kg; Plateau pressure < 28 mmHg; driving pressue < 16 cm H2O; Mechanical power < 16 Joules/min; Prevention of self-inflicted lung injury (P-SILI): ROX index > 4.8 and HACOR < 5. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with respiratory dysfunction and effective intervention / Number of patients with respiratory dysfunction X 100
Impact of standardized interventions in hemodinamic dysfunction on 48-hour delta SOFA | 48 hour
  SOSD (salvage, optimization, stabilization and de-escalation ) protocol; mean arterial pressoric taget of at least 65 mm Hg, Lactate serum level < 19 mg/dL. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hemodinamic dysfunction and effective intervention / Number of patients with hemodinamica dysfunction X 100
Impact of standardized interventions in neurologic dysfunction on 48-hour delta SOFA | 48 hour
  Image: cranial CT; Electroencephalografic monitoring and RASS Score between -1 and +1 The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with neurologic dysfunction and effective intervention / Number of patients with neurologic dysfunction X 100
Impact of standardized interventions in hematologic dysfunction on 48-hour delta SOFA | 48 hour
  Basic disease approach; avoid drugs that interfere with coagulation; Platelet transfusion in case of hemohhage; DDAVP when indicated. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hematologic dysfunction and effective intervention / Number of patients with hematologic dysfunction X 100
Impact of standardized interventions iin renal dysfunction on 48-hour delta SOFA | 48 hour
  Avoid nephotoxic drugs; Mantain mean arterial blood pressure > 65 mmHg The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with renal dysfunction and effective intervention / Number of patients with renal dysfunction X 100
Impact of standardized interventions in hepatic dysfunction on 48-hour delta SOFA | 48 hour
  Avoid hepatotoxic drugs;basic disease approach The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hepatic dysfunction and effective intervention / Number of patients with hepatic dysfunction X 100

SECONDARY OUTCOMES:
Impact of standardized interventions in respiratory dysfunction on ICU length of stay | 28 days
  Lung protective ventilation: Tidal volume 6 ml/kg; Pateau pressure < 28 mmHg; driving pressue < 16 cm H2O; Mechanical power < 16 Joules/min; Prevention of self-inflicted lung injury (P-SILI): ROX index > 4.8 and HACOR < 5. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with respiratory dysfunction and effective intervention / Number of patients with respiratory dysfunction X 100
Impact of standardized interventions in hemodinamic dysfuction on ICU length of stay | 28 days
  SOSD (salvage, optimization, stabilixation and de-escalation ) protocol; mean arterial pressoric taget of at least 65 mm Hg, Lactate serum level < 19 mg/dL. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hemodinamic dysfunction and effective intervention / Number of patients with hemodinamic dysfunction X 100
Impact of standardized interventions in neurologic dysfunction on ICU length of stay | 28 days
  Image: cranial CT; Electroencephalografic monitoring and RASS Score between -1 and +1 The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with neurologic dysfunction and effective intervention / Number of patients with neurologic dysfunction X 100
Impact of standardized interventions in hematologic dysfunction on ICU length of stay | 28 days
  Basic disease approach; avoid drugs that interfere with coagulation; Platelet transfusion in case of hemohhage; DDAVP when indicated. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hematologic dysfunction and effective intervention / Number of patients with hematologic dysfunction X 100
Impact of standardized interventions iin renal dysfunction on ICU length of stay | 28 days
  Avoid nephotoxic drugs; Mantain mean arterial blood pressure > 65 mmHg The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with renal dysfunction and effective intervention / Number of patients with renal dysfunction X 100
Impact of standardized interventions in hepatic dysfunction on ICU length of stay | 28 days
  Avoid hepatotoxic drugs;basic disease approach The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hepatic dysfunction and effective intervention / Number of patients with hepatic dysfunction X 100
Impact of standardized interventions in respiratory dysfunction on vasopressor-free days | 28 days
  Lung protective ventilation: Tidal volume 6 ml/kg; Pateau pressure < 28 mmHg; driving pressue < 16 cm H2O; Mechanical power < 16 Joules/min; Prevention of self-inflicted lung injury (P-SILI): ROX index > 4.8 and HACOR < 5. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with respiratory dysfunction and effective intervention / Number of patients with respiratory dysfunction X 100
Impact of standardized interventions in hemodinamic dysfuction on vasopressor-free days | 28 days
  SOSD (salvage, optimization, stabilixation and de-escalation ) protocol; mean arterial pressoric taget of at least 65 mm Hg, Lactate serum level < 19 mg/dL. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hemodinamic dysfunction and effective intervention / Number of patients with hemodinamic dysfunction X 100
Impact of standardized interventions in neurologic dysfunction on vasopressor-free days | 28 days
  Image: cranial CT; Electroencephalografic monitoring and RASS Score between -1 and +1 The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with neurologic dysfunction and effective intervention / Number of patients with neurologic dysfunction X 100
Impact of standardized interventions in hematologic dysfunction on vasopressor-free days | 28 days
  Basic disease approach; avoid drugs that interfere with coagulation; Platelet transfusion in case of hemohhage; DDAVP when indicated. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hematologic dysfunction and effective intervention / Number of patients with hematologic dysfunction X 100
Impact of standardized interventions iin renal dysfunction on vasopressor-free days | 28 days
  Avoid nephotoxic drugs; Mantain mean arterial blood pressure > 65 mmHg The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with renal dysfunction and effective intervention / Number of patients with renal dysfunction X 100
Impact of standardized interventions in hepatic dysfunction on vasopressor-free days | 28 days
  Avoid hepatotoxic drugs;basic disease approach The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hepatic dysfunction and effective intervention / Number of patients with hepatic dysfunction X 100
Impact of standardized interventions in respiratory dysfunction on ventilator-free days | 28 days
  Lung protective ventilation: Tidal volume 6 ml/kg; Pateau pressure < 28 mmHg; driving pressue < 16 cm H2O; Mechanical power < 16 Joules/min; Prevention of self-inflicted lung injury (P-SILI): ROX index > 4.8 and HACOR < 5. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with respiratory dysfunction and effective intervention / Number of patients with respiratory dysfunction X 100
Impact of standardized interventions in hemodinamic dysfuction on ventilator-free days | 28 days
  SOSD (salvage, optimization, stabilixation and de-escalation ) protocol; mean arterial pressoric taget of at least 65 mm Hg, Lactate serum level < 19 mg/dL. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hemodinamic dysfunction and effective intervention / Number of patients with hemodinamic dysfunction X 100
Impact of standardized interventions in neurologic dysfunction on ventilator-free days | 28 days
  Image: cranial CT; Electroencephalografic monitoring and RASS Score between -1 and +1 The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with neurologic dysfunction and effective intervention / Number of patients with neurologic dysfunction X 100
Impact of standardized interventions in hematologic dysfunction on ventilator-free days | 28 days
  Basic disease approach; avoid drugs that interfere with coagulation; Platelet transfusion in case of hemohhage; DDAVP when indicated. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hematologic dysfunction and effective intervention / Number of patients with hematologic dysfunction X 100
Impact of standardized interventions iin renal dysfunction on ventilator-free days | 28 days
  Avoid nephotoxic drugs; Mantain mean arterial blood pressure > 65 mmHg The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with renal dysfunction and effective intervention / Number of patients with renal dysfunction X 100
Impact of standardized interventions in hepatic dysfunction on ventilator-free days | 28 days
  Avoid hepatotoxic drugs;basic disease approach The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hepatic dysfunction and effective intervention / Number of patients with hepatic dysfunction X 100
Impact of standardized interventions in respiratory dysfunction on hospital length of stay | 60 days
  Lung protective ventilation: Tidal volume 6 ml/kg; Pateau pressure < 28 mmHg; driving pressue < 16 cm H2O; Mechanical power < 16 Joules/min; Prevention of self-inflicted lung injury (P-SILI): ROX index > 4.8 and HACOR < 5. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with respiratory dysfunction and effective intervention / Number of patients with respiratory dysfunction X 100
Impact of standardized interventions in hemodinamic dysfuction on hospital length of stay | 60 days
  SOSD (salvage, optimization, stabilixation and de-escalation ) protocol; mean arterial pressoric taget of at least 65 mm Hg, Lactate serum level < 19 mg/dL. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hemodinamic dysfunction and effective intervention / Number of patients with hemodinamic dysfunction X 100
Impact of standardized interventions in neurologic dysfunction on hospital length of stay | 60 days
  Image: cranial CT; Electroencephalografic monitoring and RASS Score between -1 and +1 The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with neurologic dysfunction and effective intervention / Number of patients with neurologic dysfunction X 100
Impact of standardized interventions in hematologic dysfunction on hospital length of stay | 60 days
  Basic disease approach; avoid drugs that interfere with coagulation; Platelet transfusion in case of hemohhage; DDAVP when indicated. The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hematologic dysfunction and effective intervention / Number of patients with hematologic dysfunction X 100
Impact of standardized interventions in renal dysfunction on hospital length of stay | 60 days
  Avoid nephotoxic drugs; Mantain mean arterial blood pressure > 65 mmHg The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with renal dysfunction and effective intervention / Number of patients with renal dysfunction X 100
Impact of standardized interventions in hepatic dysfunction on hospital length of stay | 60 days
  Avoid hepatotoxic drugs;basic disease approach The effectiveness of the interventions on organic disfunction will be evaluated through the formula:
  Number of patients with hepatic dysfunction and effective intervention / Number of patients with hepatic dysfunction X 100

CONTACTS AND LOCATIONS:
Overall Officials: JOSE R AZEVEDO, MD, PhD, Study Director — Hospital Sao Domingos; BARBARA L RIBEIRO, MD, Principal Investigator — Hospital Sao Domingos
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anami EH, Grion CM, Cardoso LT, Kauss IA, Thomazini MC, Zampa HB, Bonametti AM, Matsuo T. Serial evaluation of SOFA score in a Brazilian teaching hospital. Intensive Crit Care Nurs. 2010 Apr;26(2):75-82. doi: 10.1016/j.iccn.2009.10.005. Epub 2009 Dec 29. PMID 20036543
- [Result] Bone RC, Sibbald WJ, Sprung CL. The ACCP-SCCM consensus conference on sepsis and organ failure. Chest. 1992 Jun;101(6):1481-3. doi: 10.1378/chest.101.6.1481. No abstract available. PMID 1600757
- [Result] Moreno R, Vincent JL, Matos R, Mendonca A, Cantraine F, Thijs L, Takala J, Sprung C, Antonelli M, Bruining H, Willatts S. The use of maximum SOFA score to quantify organ dysfunction/failure in intensive care. Results of a prospective, multicentre study. Working Group on Sepsis related Problems of the ESICM. Intensive Care Med. 1999 Jul;25(7):686-96. doi: 10.1007/s001340050931. PMID 10470572
- [Result] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Result] Jones AE, Trzeciak S, Kline JA. The Sequential Organ Failure Assessment score for predicting outcome in patients with severe sepsis and evidence of hypoperfusion at the time of emergency department presentation. Crit Care Med. 2009 May;37(5):1649-54. doi: 10.1097/CCM.0b013e31819def97. PMID 19325482
- [Result] de Azevedo JR, Torres OJ, Beraldi RA, Ribas CA, Malafaia O. Prognostic evaluation of severe sepsis and septic shock: procalcitonin clearance vs Delta Sequential Organ Failure Assessment. J Crit Care. 2015 Feb;30(1):219.e9-12. doi: 10.1016/j.jcrc.2014.08.018. Epub 2014 Sep 10. PMID 25241933
- [Result] Soo A, Zuege DJ, Fick GH, Niven DJ, Berthiaume LR, Stelfox HT, Doig CJ. Describing organ dysfunction in the intensive care unit: a cohort study of 20,000 patients. Crit Care. 2019 May 23;23(1):186. doi: 10.1186/s13054-019-2459-9. PMID 31122276
- [Result] de Grooth HJ, Geenen IL, Girbes AR, Vincent JL, Parienti JJ, Oudemans-van Straaten HM. SOFA and mortality endpoints in randomized controlled trials: a systematic review and meta-regression analysis. Crit Care. 2017 Feb 24;21(1):38. doi: 10.1186/s13054-017-1609-1. PMID 28231816